CLINICAL TRIAL: NCT07124936
Title: A Phase 1b/2 Study to Evaluate the Safety, Tolerability, and Antitumor Activity of HDM2005 in Combination With Standard of Care in Patients With Diffuse Large B-Cell Lymphoma
Brief Title: A Study of HDM2005 in Combination With Standard of Care in Patients With Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDM2005-104
Record Dates: First submitted 2025-08-11; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Gemcitabine; Oxaliplatin; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with r/r DLBCL (Cohort A) (Experimental): Participants with r/r DLBCL will receive a dose of HDM2005 (1.8 mg/kg or 2.0 mg/kg, on Day 2 Cycle 1 and Day 1 Cycle 2 to 6-8) plus 1000 mg/ m^2 gemcitabine (on Day 2 Cycle 1 and Day 1 Cycle 2 to 6-8), 100 mg/ m^2 oxaliplatin, and 375 mg/m^2 rituximab or rituximab biosimilar administered by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 6-8 cycles.
  Interventions: Drug: HDM2005; Drug: Rituximab or Rituximab biosimilar; Drug: Gemcitabine; Drug: Oxaliplatin
- Participants with untreated DLBCL (Cohort B) (Experimental): Participants with untreated DLBCL will receive a dose of HDM2005 (1.8 mg/kg or 2.0 mg/kg, on Day 2 Cycle 1 and Day 1 Cycle 2 to 6) plus 750 mg/m^2 cyclophosphamide (on Day 2 Cycle 1 and Day 1 Cycle 2 to 6), 50 mg/m^2 doxorubicin (on Day 2 Cycle 1 and Day 1 Cycle 2 to 6), and 375 mg/m^2 rituximab or rituximab biosimilar administered by intravenous (IV) infusion on Day 1 and 2 Cycle 1 and Day 1 Cycle 2 to 6 of each 3-week cycle for up to 6 cycles. Participants will also receive 100 mg prednisone or prednisolone via oral tablet per day during Days 1-5 of each 3-week cycle for up to 6 cycles.
  Interventions: Drug: HDM2005; Drug: Rituximab or Rituximab biosimilar; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: HDM2005 — HDM2005 will be administered as an intravenous injection.
Drug: Rituximab or Rituximab biosimilar — Rituximab or Rituximab biosimilar will be administered as an intravenous injection.
Drug: Gemcitabine — Gemcitabine will be administered as an intravenous injection.
  Arms: Participants with r/r DLBCL (Cohort A)
Drug: Oxaliplatin — Oxaliplatin will be administered as an intravenous injection.
  Arms: Participants with r/r DLBCL (Cohort A)
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an intravenous injection.
  Arms: Participants with untreated DLBCL (Cohort B)
Drug: Doxorubicin — Doxorubicin will be administered as an intravenous injection.
  Arms: Participants with untreated DLBCL (Cohort B)
Drug: Prednisone — Prednisone will be administered orally.
  Arms: Participants with untreated DLBCL (Cohort B)

SUMMARY:
The purpose of this phase 1b/2 study is to evaluate the safety, tolerability, and antitumor activity of HDM2005 in combination with standard of care in participants with diffuse large B-cell lymphoma. This study will include two arms: Cohort A (HDM2005 + R-GemOx) will enroll participants with relapsed/refractory DLBCL. Cohort B (HDM2005 + R-CHP) will enroll participants with untreated DLBCL. The study will consist of two parts: dose-escalation part and dose-expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Life expectancy >12 weeks.
4. Histologically confirmed diffuse large B-cell lymphoma (DLBCL).

   a. Cohort B: International Prognostic Index (IPI) score of 2-5.
5. Prior treatment:

   1. Cohort A: At least one (≥1) line of prior systemic therapy.
   2. Cohort B: Has received no prior treatment for DLBCL.
6. At least one bi-dimensionally measurable (≥1.5 cm) nodal lesion, or one bi-dimensionally measurable (≥1 cm) extranodal lesion, as measured on computed tomography (CT) scan.
7. Adequate organ system and hematologic function as defined in protocol.

Exclusion Criteria:

1. Known active central nervous system (CNS) lymphoma.
2. Prior of allogeneic hematopoietic stem cell transplantation and has acute or ongoing graft-versus-host disease (GVHD) of any grade.
3. Known additional malignancy that is progressing or has required active treatment within the past 3 years.
4. History of severe bleeding disorders.
5. History of interstitial lung disease or radiation pneumonitis.
6. Prior solid organ transplant.
7. Ongoing Grade >1 treatment-related adverse events.
8. Current or history of clinically significant cardiovascular and cerebrovascular diseases.
9. Active infection requiring systemic therapy.
10. Concurrent active HBV or HCV infection or known history of human immunodeficiency virus (HIV) infection.
11. Prior ROR1-targeted therapy.
12. Ongoing corticosteroid therapy.
13. Current active autoimmune disease or history of autoimmune disease requiring treatment.
14. History of drug anaphylaxis or severe food allergy.
15. Any history or current evidence of disease, treatment, or laboratory abnormality as determined by the investigator that may affect the study results, interfere with the subject's full participation in the study, or be contrary to the subject's best interests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-10-26 (Estimated); Study Completion 2029-10-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience dose-limiting toxicities (DLTs) in dose-escalation part | Up to ~3 weeks
  The CTCAE, Version 5.0 will be used to grade the severity of AEs in this study. DLTs will be reported for dose-escalation part of this study.
Number of participants who experience adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) in dose-escalation part | Up to ~54 months
  Incidence and grading of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) (based on the National Cancer Institute's Common Terminology Criteria for Adverse Events [CTCAE] version 5.0). Incidence of treatment interruption and dose adjustment due to AEs and changes in laboratory tests, vital signs, physical examination, electrocardiogram (ECG), and Eastern Cooperative Oncology Group (ECOG) performance status score.
Complete response (CR) rate in dose-expansion part | Up to ~30 months
  CR rate is defined as the percentage of participants who achieve a complete response (CR) per Lugano criteria, as determined by the investigator
RP2D of HDM2005 | Up to ~30 months
  Recommended phase 2 dose of HDM2005 in combination with SoC in patients with r/r DLBCL and untreated DLBCL

SECONDARY OUTCOMES:
Plasma concentration of HDM2005, total antibody and monomethyl auristatin E (MMAE) | Up to ~30 months
  Plasma concentration of HDM2005, total antibody and MMAE will be reported for each dose level
Number of participants positive for anti-drug antibodies (ADA) | Up to ~30 months
  Number of participants with positive ADA will be assessed
Number of participants who experience adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) in dose-expansion part | Up to ~54 months
  Incidence and grading of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) (based on the National Cancer Institute's Common Terminology Criteria for Adverse Events [CTCAE] version 5.0). Incidence of treatment interruption and dose adjustment due to AEs and changes in laboratory tests, vital signs, physical examination, electrocardiogram (ECG), and Eastern Cooperative Oncology Group (ECOG) performance status score.
Objective response rate (ORR) | Up to ~30 months
  ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per Lugano criteria as determined by the investigator
Progression-free survival (PFS) | Up to ~54 months
  PFS is defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression/relapse or death from any cause, whichever occurs first as determined by the investigator
Duration of response (DOR) | Up to ~54 months
  DOR is defined as the interval from the first documentation of CR or PR until disease progression or death due to any cause, whichever occurs first
Time to response (TTR) | Up to ~54 months
  TTR is defined as the interval from the start of study therapy to the first documentation of CR or PR
Time to progression (TTP) | Up to ~54 months
  TTP is defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression as determined by the investigator
Overall survival (OS) | Up to ~54 months
  OS is defined as the time from randomization to death due to any cause

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - HunanCancer Hospital, Changsha, Hunan
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute,Shandong Cancer Hospital), Jinan, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Kunming Medical UniversityThe Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided